CLINICAL TRIAL: NCT05995184
Title: Association Between Metacognitive Awareness of Pediatric Nursing Students and Their Academic Achievement: A Correletional Study
Brief Title: Metacognitive Awareness, Pediatric Nursing, Students, Academic Achievement
Status: Completed | Type: Observational
Sponsor: Matrouh University (Other)
Collaborators: Damnhour University (Unknown)
Responsible Party: Principal Investigator, Seham El-Sayed Saleh Hassan, Lecturer of pediatric nursing, faculty of nursing, Matrouh University
Other Study IDs: 68-a (15/12/2022)
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Achievement
Keywords: 1 - Metacognitive Awareness; 2 - Pediatric Nursing; 3 - Students Achievement

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
* Metacognitive Awareness
* Pediatric Nursing
* Students Achievement

DETAILED DESCRIPTION:
* The study was carried out at Faculty of Nursing Damanhour University Egypt. The Faculty of Nursing has nine different scientific nursing departments including pediatric nursing department. Pediatric nursing is one of the main courses was taught for the students enrolled in the third year in each term in the third scholastic year. Each term is consisting of 15 weeks. The clinical training (rotation) is given 12 hours /week.
* The present study subjects comprised of 150 students. The sample size was determined by using EPI Info 7 program using the following information: Population size = 500 (total no. of pediatric nursing students during the 2nd term of the academic year 2022 -2023), expected frequency =50%, acceptable error= 10%, confidence coefficient = 99%, which revealed a simple size = 125.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric nursing students
* Third year
* 19-23 years

Exclusion Criteria:

* None

Ages: 19 Years to 23 Years | Sex: All
Age Groups: Adult
Study Population: Pediatric nursing students =500 divided into 10 equal groups. The study subjects were randomly selected using simple random sampling technique 15students from each group. The total sample size is 150 students.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2023-02-25 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
The Pediatric Nursing Achievement tool | three months
  It was developed by the researchers guided by the Pediatric Nursing notes that was developed by the Pediatric Nursing Staff of the Faculty of Nursing Damanhour University (2020)
Metacognitive Awareness Inventory | three months
  It consisted of 52 items divided into two broad parts; the first part: Knowledge about cognition (17 items). The second part: Regulation of cognition (35 items)

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Damnhour University, Damnhour
  - Matrouh university, Marsá Maţrūḩ

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] (1) Metacognition and Problem-Solving Strategies Feral Ogan- BekirogluMarmara UniversityZeynep DulgerMarmara University, by F Ogan-Bekiroglu - Swanson, H. L. (1990). Influence of Metacognitive knowledge and aptitude on problem solving. Journal of Educafional Psychology, 82(2), 306-314. 6 pages•1
- [Background] Li S, de Ala M, Mao D, Wang A, Wu C. Effect of a Nursing Comprehensive Skill Training Course (NCST-C) on Nursing Students' Metacognitive Awareness: A Quasi-experimental Study. Asian Nurs Res (Korean Soc Nurs Sci). 2022 Dec;16(5):275-281. doi: 10.1016/j.anr.2022.10.003. Epub 2022 Nov 1. PMID 36332792
- [Background] Asadzandi S, Mojtahedzadeh R, Mohammadi A. What are the Factors that Enhance Metacognitive Skills in Nursing Students? A Systematic Review. Iran J Nurs Midwifery Res. 2022 Nov 18;27(6):475-484. doi: 10.4103/ijnmr.ijnmr_247_21. eCollection 2022 Nov-Dec. PMID 36712305
- [Background] Metacognition and Problem-Solving Strategies Feral Ogan- BekirogluMarmara UniversityZeynep DulgerMarmara University, by F Ogan-Bekiroglu - Swanson, H. L. (1990). Influence of Metacognitive knowledge and aptitude on problem solving. Journal of Educafional Psychology, 82(2), 306-314. 6 pages•1
- [Background] Salari M., Rohaniahmad T, Ramlah H, Zarida H. Meta-Cognitive Strategies and Nursing Students' Achievement. Yasuj University of Medical Sciences, Yasuj, Journal of Education and Vocational Research, Vol. 4, No. 6, pp. 169-173, June 2013 (ISSN 2221-2590).
- [Background] Medina MS, Castleberry AN, Persky AM. Strategies for Improving Learner Metacognition in Health Professional Education. Am J Pharm Educ. 2017 May;81(4):78. doi: 10.5688/ajpe81478. PMID 28630519